CLINICAL TRIAL: NCT06229275
Title: A Study to Evaluate the Effectiveness of the Rover Cervex-Brush Device vs. the Personal Pap Smear Device™ for Collection of Cervical Cells for Detecting Cervical Dysplasia or Neoplasia
Brief Title: Comparing Effectiveness of Physician-assisted Versus Self-assisted Pap Smear Collection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Morehouse School of Medicine (Other)
Collaborators: GyneConcepts, Inc. (Unknown)
Responsible Party: Principal Investigator, Regina Leonis, Assistant Professor, Morehouse School of Medicine
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: 2011440
Record Dates: First submitted 2024-01-10; First posted 2024-01-29 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Cervical Cancer Screening
Keywords: pap smear collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Pap smear collection using the Personal Pap Smear (PPS) Device (Experimental): The investigational device, trade named the Personal Pap Smear™ (PPS) developed by GyneConcepts of Atlanta, Georgia. It arrives completely assembled, and ready-for-use, in a sealed plastic bag. The PPS device is a multi-component assembly designed for the collection of exfoliated cervical epithelial cells. Its four major components are the (1) Tube Body, (2) U-Ring and attached Aligning Spoon, (3) Ball Handle, (with permanently anchored bristle Collection Brush), and (4) Safety Cover.
  Interventions: Device: Pap smear collection using the Personal Pap Smear (PPS) Device
- Pap smear collection using the Rovers Cervex-Brush (Active Comparator): The Predicate device utilized in this study is the Cervix-Examination Brush, manufactured by Rover (Manufacturers Code: 9443). The Cervex-Brush (CervixExamination Brush) is made of polyethylene and has a total length of 20 centimeters. The top portion uses a soft flexible brush to obtain cell samples. The brush consists of 57 semi-circular plastic bristles of various lengths. The shape is such that the top edges of the brush follow the contours of the cervix. The longer middle bristles reach deep into the endocervical canal- 'Os'. The shorter bristles touch both the ectocervical area and transformation zone at the same time. This device is packaged with identical standards used for packaging commercial tampons.
  Interventions: Device: Active Comparator: Pap smear collection using the Rovers Cervex-Brush

INTERVENTIONS:
Device: Pap smear collection using the Personal Pap Smear (PPS) Device — Diagnostic Test: Use of PPS device to collect cervical cells during pap smear collection.
  Arms: Pap smear collection using the Personal Pap Smear (PPS) Device
Device: Active Comparator: Pap smear collection using the Rovers Cervex-Brush — Diagnostic Test: Use of Rovers Cervex-Brush to collect cervical cells during pap smear collection.
  Arms: Pap smear collection using the Rovers Cervex-Brush

SUMMARY:
This purpose of this research study is to determine the effectiveness of the Personal Pap Smear Device™ to collect adequate cervical cell samples for cytology examination when compared with the Rover Cervex-Brush (Cervix-Examination Brush).

DETAILED DESCRIPTION:
To determine the effectiveness of the Personal Pap Smear Device™ to collect adequate (as defined by Bethesda Guidelines 2014) cervical cell samples for cytology examination as compared with the Rover Cervex-Brush (Cervix-Examination Brush).

ELIGIBILITY:
Inclusion Criteria:

* Adult women, aged 21-65 years old.
* Do not have any medical or psychiatric condition affecting the ability to give voluntary informed consent.
* Be able to read and understand English

Exclusion Criteria:

* Participants currently on menses
* Inability to provide Informed Consent
* Previous total hysterectomy
* History of radiation treatment for cervical cancer
* Pregnancy
* Medical condition that interferes with conduct of study, in investigator's opinion
* Evidence of active cervical infection requiring treatment
* Known bleeding diathesis

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of the samples for the Predicate Device versus PPS device | Baseline
  Data of Adequate versus Inadequate will be reported to include a positive percent agreement (PPA) defined as PPA= A/(A+C) and the negative percent agreement (NPA) defined as NPA = D/(B+D) along with their 95% confidence bounds using the Clopper-Pearson method.

SECONDARY OUTCOMES:
The Comparison of Cell Types of the PPS Device versus the Predicate Device | Baseline
  The PPS Device and the Predicate Device cell types will be measured against the 2014 Bethesda cytology categories that will be displayed in a 8 x 8 contingency table.

CONTACTS AND LOCATIONS:
Overall Officials: Regina K Leonis, MD, MD, Principal Investigator — Morehouse School of Medicine
Locations (1):
- Morehouse School of Medicine, Atlanta, Georgia, United States